CLINICAL TRIAL: NCT02382003
Title: Testing Target Engagement and Effectiveness of Web-based Interpretation Training For Anxiety
Brief Title: Web-based Interpretation Training For Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bethany A. Teachman, Ph.D., Professor, Department of Psychology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0331-00
Record Dates: First submitted 2015-02-16; First posted 2015-03-06 (Estimated); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Anxiety
Keywords: Anxiety; Cognitive bias; Telemedicine
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Positive Training+Anxious Imagery Prime (Experimental): Positive Cognitive Bias Modification - Interpretation training paired with a preceding Anxious Imagery Prime
  Interventions: Behavioral: Positive Cognitive Bias Modification - Interpretation; Behavioral: Anxious Imagery Prime
- Positive Training+Neutral Imagery Prime (Experimental): Positive Cognitive Bias Modification - Interpretation training paired with a preceding Neutral Imagery Prime
  Interventions: Behavioral: Positive Cognitive Bias Modification - Interpretation; Behavioral: Neutral Imagery Prime
- 50/50 Training+Anxious Imagery Prime (Active Comparator): 50/50 Cognitive Bias Modification - Interpretation (half positive & half negative scenarios) paired with a preceding Anxious Imagery Prime
  Interventions: Behavioral: 50/50 Cognitive Bias Modification - Interpretation; Behavioral: Anxious Imagery Prime
- 50/50 Training+Neutral Imagery Prime (Active Comparator): 50/50 Cognitive Bias Modification - Interpretation (half positive & half negative scenarios) paired with a preceding Neutral Imagery Prime
  Interventions: Behavioral: 50/50 Cognitive Bias Modification - Interpretation; Behavioral: Neutral Imagery Prime
- No Scenario+Anxious Imagery Prime (Other): No scenarios paired with a preceding Anxious Imagery Prime
  Interventions: Behavioral: Anxious Imagery Prime
- No Scenario+Neutral Imagery Prime (Other): No scenarios paired with a preceding Neutral Imagery Prime
  Interventions: Behavioral: Neutral Imagery Prime

INTERVENTIONS:
Behavioral: Positive Cognitive Bias Modification - Interpretation — Training involves presenting participants with brief scenarios that introduce an ambiguous potential threat. Critically, the ambiguity regarding how the situation is resolved remains until the last word of the scenario, which is presented as a word fragment that the participant must solve, which will then assign a benign (rather than threatening) meaning to the scenario.
  Other Names: Ambiguous Scenarios Training
  Arms: Positive Training+Anxious Imagery Prime; Positive Training+Neutral Imagery Prime
Behavioral: 50/50 Cognitive Bias Modification - Interpretation — This condition follows the same design and content as the Positive Training conditions, except the word fragments differ; rather than consistently resolving the scenario in a positive direction, half of the scenarios will end with a negative (anxiety-congruent) word fragment, and half will end with a positive word fragment.
  Arms: 50/50 Training+Anxious Imagery Prime; 50/50 Training+Neutral Imagery Prime
Behavioral: Anxious Imagery Prime — We will test whether priming anxious concerns and feared negative outcomes on the web via the addition of a guided anxious imagery prime at the start of each session will enhance effects.
  Arms: 50/50 Training+Anxious Imagery Prime; No Scenario+Anxious Imagery Prime; Positive Training+Anxious Imagery Prime
Behavioral: Neutral Imagery Prime — At the start of each session, participants will complete a neutral control imagery exercise where they do a guided imagery exercise imagining upcoming mundane tasks, like brushing one's teeth.
  Arms: 50/50 Training+Neutral Imagery Prime; No Scenario+Neutral Imagery Prime; Positive Training+Neutral Imagery Prime

SUMMARY:
The study aims to develop a web-based Cognitive Bias Modification infrastructure to train interpretations, and evaluate the usability, acceptability, and feasibility of the program to reduce anxiety symptoms.

DETAILED DESCRIPTION:
Approximately half of the U.S. population experiences serious mental health problems during their lifetime, including 29% with anxiety pathology severe enough to qualify for an anxiety disorder diagnosis [1]. Critically, more than two thirds of individuals struggling with a mental illness do not receive treatment [1]. With this level of mental illness burden, it is clear that treating people one-on-one in an office setting will never meet the existing needs [2]. There are many barriers to treatment, including costs [3], difficulties accessing evidence-based treatments in many regions [4], and associated stigma [5]. Thus, there is a pressing need to consider alternative, larger scale approaches to delivering mental health services. Cognitive Bias Modification (CBM) interventions hold considerable promise as a way to meet these needs, especially for anxiety difficulties [6]. These computer-based programs are designed to alter biased ways of thinking, such as a tendency toward negative interpretations, which cause and maintain anxiety [6]. Because these programs do not require therapist contact and can be administered on any computer with an Internet connection, CBM holds promise as a cost-effective method that can be disseminated widely. However, while CBM for interpretation bias (CBM-I) has established efficacy when administered in-person in the laboratory [7], it now needs to be tested with broader populations using a web-based infrastructure to examine: a) whether the program will be effective in a web environment, b) whether the program continues to engage the targeted mechanism (i.e., interpretation bias), c) the feasibility of this delivery method, and d) the modifications needed to adapt the program for the web (in particular, to prime anxiety-linked negative thinking in an online environment, we test the effect of adding a guided anxious imagery exercise to prime feared outcomes prior to each training session).

Together, the current proposal will develop an infrastructure to pilot test the effectiveness of web-based CBM-I for anxiety symptoms. CBM-I training will target moderate to severe anxiety symptoms, a widespread problem area with considerable occupational and social impairment [8]. Participants will be visitors to Project Implicit Mental Health (PIMH), an existing website directed by the Principal Investigator that allows visitors to assess their cognitive biases tied to mental health concerns. Consistent with the RFA's priorities, this approach encourages efficiencies by capitalizing on the existing PIMH site and its heavy traffic. Further, the site's large number of visitors and use of automated assessments will make it efficient to assess baseline demographic characteristics and interpretation bias as moderators of CBM-I effects that can be tested in future trials.

Aim 1: Develop and evaluate usability and acceptability of web-based CBM-I for anxiety symptoms.

Aim 1 will build the web-based interpretation bias training program using the PIMH infrastructure. We will pilot the program on a small test group of moderate to highly anxious participants (N=15) who will complete questionnaires and semi-structured interviews to provide feedback on the programs' usability and acceptability. Further, an advisory board (N=8) of anxiety researchers, clinicians, and experts in CBM and web-based research will provide feedback on the program and study protocol. Using a "deployment-focused" approach, this feedback from experts and end-users will be used to iteratively modify the program for the trial planned for Aims 2 and 3. Thus, even at this initial pilot stage, we will measure the targeted outcome (anxiety symptoms) and mechanism (interpretation bias) to determine whether modifications to enhance target engagement are needed. Note, within Research Domain Criteria (RDoC), this outcome falls under the Potential Threat/Anxiety construct within the Negative Valence System, and the targeted mechanism (interpretation bias) falls under the Response Selection, Inhibition construct within the Cognitive (effortful) control system. Both the outcome and mechanism will be objectively measured using multiple units of analysis (e.g., behavior and self-report). Further, mechanisms underlying the guided anxious imagery prime's effects will be measured by assessing subjective distress, imagery vividness, and activation of feared outcomes following the manipulation. This prime was selected in part because of its potential to be disseminated widely in future trials, given it does not require human contact.

Aim 2: Test target engagement, feasibility and effectiveness of web-based CBM-I.

Aim 3: Evaluate the impact of an anxious prime on web-based CBM-I for anxiety symptoms.

Aims 2 and 3 will test the feasibility of an 8-session web-based interpretation training program among individuals with moderate to severe anxiety symptoms (based on screening at the PIMH site). Participants will be randomly assigned to positive CBM-I (90% positive scenario training), 50% positive/50% negative CBM-I, or a no scenario control condition. Half the participants in each of these 3 conditions will receive an anxious imagery prime prior to each training session, and half will receive a neutral imagery prime, resulting in a 3 training condition x 2 prime design (N=210; target of n=35 per condition). Feasibility will be determined by analyses of recruitment, attrition, acceptance of randomization, adherence to and appropriateness of the measurement model, caseness, extent of missing data, and safety. Additionally, target engagement (change in interpretation bias) and preliminary tests of effectiveness at reducing anxiety symptoms will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

The target population will be adults age 18 and over who score in the moderate to extremely severe anxiety range (i.e., 10 or higher) on the Depression, Anxiety, Stress Scales - Short Form: Anxiety Subscale and have regular access to the Internet.

Exclusion Criteria:

None listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 807 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Teachman, PhD, Principal Investigator — University of Virginia
Locations (1):
- MindTrails web site: https://mindtrails.virginia.edu/ (thru Univ. of Virginia), Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Steinman SA, Portnow S, Billingsley AL, Zhang D, Teachman BA. Threat and benign interpretation bias might not be a unidimensional construct. Cogn Emot. 2020 Jun;34(4):783-792. doi: 10.1080/02699931.2019.1682973. Epub 2019 Oct 25. PMID 31650889

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Started | 111 | 141 | 121 | 144 | 136 | 154
Completed (We marked participants as "completed" if they made it to session 6 due to attrition.) | 10 | 25 | 13 | 22 | 13 | 22
Not Completed | 101 | 116 | 108 | 122 | 123 | 132

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime | Total
Number analyzed (Participants) | 111 | 141 | 121 | 144 | 136 | 154 | 807
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.42 (13.04) | 32.22 (12.22) | 32.06 (12.39) | 34.22 (14.51) | 33.45 (13.37) | 35.16 (14.39) | 33.59 (13.32)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender (Female) | 79 | 106 | 87 | 104 | 94 | 113 | 583
  Male | 31 | 31 | 29 | 38 | 37 | 37 | 203
  Other | 1 | 2 | 1 | 1 | 1 | 2 | 8
  Prefer not to answer | 0 | 1 | 2 | 0 | 2 | 1 | 6
  Transgender | 0 | 1 | 1 | 1 | 2 | 1 | 6
  Not reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/European Origin | 85 | 116 | 92 | 109 | 103 | 121 | 626
  Black/African Origin | 5 | 2 | 3 | 5 | 5 | 4 | 24
  East/South Asian | 8 | 11 | 7 | 15 | 12 | 10 | 63
  American Indian/Alaska Native | 2 | 0 | 2 | 0 | 2 | 0 | 6
  Other or Unknown | 8 | 5 | 8 | 10 | 10 | 13 | 54
  Prefer not to answer | 3 | 6 | 7 | 5 | 4 | 5 | 30
  Not reported | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian/Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic/Latino | 89 | 115 | 108 | 108 | 115 | 132 | 667
  Hispanic/Latino | 11 | 11 | 5 | 17 | 13 | 10 | 67
  Prefer not to answer | 4 | 9 | 5 | 11 | 6 | 6 | 41
  Unknown | 7 | 5 | 2 | 8 | 2 | 5 | 29
  Not reported | 0 | 1 | 1 | 0 | 0 | 1 | 3
Marital Status [Count of Participants; unit: Participants]
  Married | 40 | 40 | 28 | 42 | 45 | 52 | 247
  Single | 28 | 47 | 47 | 51 | 42 | 50 | 265
  Prefer not to answer | 1 | 3 | 3 | 2 | 0 | 4 | 13
  Other options | 42 | 51 | 43 | 49 | 49 | 48 | 282
Education [Count of Participants; unit: Participants]
  High school or below | 8 | 10 | 15 | 11 | 11 | 12 | 67
  Graduate school | 34 | 33 | 32 | 46 | 44 | 47 | 236
  Bachelor's degree | 33 | 38 | 27 | 34 | 29 | 39 | 200
  Other | 36 | 59 | 46 | 53 | 52 | 56 | 302
  Not reported | 0 | 1 | 1 | 0 | 0 | 0 | 2
Income [Count of Participants; unit: Participants]
  < $75,000 | 49 | 66 | 53 | 54 | 56 | 72 | 350
  > $200,000 | 5 | 5 | 5 | 7 | 9 | 4 | 35
  Between $75,000 and $200,000 | 38 | 37 | 36 | 47 | 38 | 47 | 243
  Prefer not to answer | 9 | 20 | 15 | 19 | 19 | 15 | 97
  Not reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Don't know | 10 | 12 | 12 | 17 | 14 | 16 | 81
Employment Status [Count of Participants; unit: Participants]
  Working full-time | 56 | 52 | 41 | 62 | 54 | 72 | 337
  Student | 31 | 46 | 36 | 41 | 37 | 38 | 229
  Working part-time | 12 | 15 | 25 | 15 | 11 | 13 | 91
  Unemployed or looking for work | 6 | 9 | 7 | 9 | 15 | 11 | 57
  Retired | 2 | 4 | 2 | 5 | 4 | 9 | 26
  Other | 4 | 14 | 9 | 12 | 13 | 11 | 63
  Not reported | 0 | 1 | 1 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Recognition Ratings (Positive Interpretation Bias)
Description: To measure interpretation bias, participants will read ambiguous scenarios with titles, after which they will see the titles of each scenario, followed by 2 disambiguated interpretations of the scenario: 1 positive and 1 negative. Participants will rate each disambiguated interpretation based on how similar in meaning it is to the original scenario on a 4-point scale ranging from 1 to 4. The mean of the positive, threat-related ratings index positive interpretation bias. Higher scores represent a more positive interpretation bias.
Time Frame: Baseline, and after sessions 3 (~2 weeks following baseline), 6 (~10 days after session 3), and 8 (~7 days after session 6) & at 2-month follow-up. Measure will be completed immediately following that day's training session.
Population: Due to attrition, the number of participants differs at each session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 111 | 141 | 121 | 144 | 136 | 154
score on a scale
  Baseline: number analyzed (Participants) | 110 | 140 | 120 | 143 | 110 | 125
  Baseline | 1.23 (0.87) | 1.19 (0.82) | 1.22 (0.83) | 1.16 (0.88) | 1.17 (0.83) | 1.22 (0.83)
  Session 3: number analyzed (Participants) | 23 | 41 | 25 | 40 | 32 | 47
  Session 3 | 1.63 (0.90) | 1.57 (0.83) | 1.47 (0.70) | 1.38 (0.94) | 1.20 (0.77) | 1.43 (0.71)
  Session 6: number analyzed (Participants) | 15 | 28 | 15 | 22 | 13 | 25
  Session 6 | 1.67 (0.78) | 1.47 (0.79) | 1.50 (0.85) | 1.30 (0.98) | 1.33 (0.82) | 1.51 (0.71)
  Session 8: number analyzed (Participants) | 9 | 22 | 10 | 20 | 12 | 14
  Session 8 | 1.58 (0.78) | 1.38 (0.74) | 1.72 (0.76) | 1.43 (0.97) | 1.42 (0.63) | 1.38 (0.66)
  2-month Follow-up: number analyzed (Participants) | 2 | 4 | 4 | 5 | 7 | 2
  2-month Follow-up | 1.50 (1.16) | 1.64 (0.51) | 1.47 (0.81) | 1.24 (0.73) | 1.62 (0.68) | 2.05 (0.79)
Statistical Analysis 1: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; Effect of CBM-I condition: The main effect of CBM-I was represented by three binary variables in the main effect models (Positive vs. No-training control; 50/50 vs. No- training control; Positive vs. 50/50). Due to high attrition, latent growth curve modeling was used instead of the planned approach (mixed effects models with multiple imputation of missing values) to minimize bias due to missing data estimation. Because omnibus tests were not run, results for all comparisons are listed below; Test type: Superiority; p = 0.005, Likelihood Ratio Tests — =Positive~No-training, 0.030=Positive~50/50 training, 0.833=50/50~No-training Alpha = .05; 2=df Positive~No-training, 2=df Positive~50/50 training, 2=df 50/50~No-training; Mean Difference (Net) = 10.730 — =Positive~No-training, 7.053=Positive~50/50 training, 0.366=50/50~No-training
Statistical Analysis 2: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; Effect of Imagery Prime Type: The main effect of imagery prime was represented by one binary variable (neutral vs. anxiety imagery). Due to high attrition, latent growth curve modeling was used instead of the planned approach (mixed effects models with multiple imputation of missing values) to minimize bias due to missing data estimation. Because omnibus tests were not run, results for all comparisons are listed below; Test type: Superiority; p = 0.799, Likelihood Ratio Tests — =Neutral~Anxiety prime Alpha = .05; 2=df Neutral~Anxiety prime; Mean Difference (Net) = 0.449 — =Neutral~Anxiety prime
Statistical Analysis 3: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; Effect of CBM-I condition and Imagery Prime Type interaction: Each cell of the interaction was represented by one of 5 binary variables, set to 1 if a participant was in that group, and 0 otherwise; the sixth group (No-training + neutral prime) was considered a reference group, and was represented by all variables being 0. Due to high attrition, latent growth curve modeling was used instead of the planned approach. Because omnibus tests were not run, results for all comparisons are listed below; Test type: Superiority; p = 0.011, Likelihood Ratio Tests — =No-train+Neut~Pos+Anx, 0.026=No-train+Neut~Pos+Neut, 0.094=No-train+Anx~Pos+Anx, 0.170=No-train+Anx~Pos+Neut, No-train(all)~50/50(all)≥ 0.136; 2=all df; Mean Difference (Net) = 9.085 — =No-train+Neut~Pos+Anx, 7.328=No-train+Neut~Pos+Neut, 4.722=No-train+Anx~Pos+Anx, 3.547=No-train+Anx~Pos+Neut, No-train(all)~50/50(all)≤3.988

2. Primary Outcome: Change in Overall Anxiety Severity and Impairment Scale
Description: The Overall Anxiety Severity and Impairment Scale (OASIS; Norman, Hami Cissell, Means-Christensen, & Stein, 2006) assesses anxiety frequency, severity, and associated avoidance, work and social interference. This 5-item measure of anxiety symptom severity and impairment has good psychometric properties, shows treatment sensitivity, and is valid in community and clinical samples. All items are rated on a scale of 0 (lowest impairment/severity) to 4 (highest impairment/severity). Total scores on the OASIS are calculated by summing the scores of each of the 5 questions. The total score on the OASIS ranges from 0 to 20, with higher scores indicating greater anxiety. A cut-score of 8 or higher on the OASIS is considered to indicate probable anxiety disorder.
Time Frame: Baseline, and after sessions 1,2,3,4,5,6,7,8 (sessions will be spaced ~3-4 days apart) & at 2-month follow-up. Measure will be completed immediately following that day's training session. Session 2 is expected to occur within 3-8 days of the baseline.
Population: Due to attrition, the number of participants differs at each session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 111 | 141 | 121 | 144 | 136 | 154
score on a scale
  Baseline: number analyzed (Participants) | 106 | 135 | 117 | 136 | 129 | 144
  Baseline | 10.367925 (0.65) | 11.066667 (0.63) | 11.470085 (0.62) | 10.544118 (0.69) | 11.131783 (0.60) | 10.486111 (0.67)
  Session 1: number analyzed (Participants) | 72 | 96 | 83 | 90 | 92 | 103
  Session 1 | 10.152778 (0.55) | 10.458333 (0.60) | 11.168675 (0.58) | 10.011111 (0.58) | 10.836957 (0.55) | 10.271845 (0.63)
  Session 2: number analyzed (Participants) | 51 | 63 | 53 | 70 | 81 | 96
  Session 2 | 8.725490 (0.57) | 9.587302 (0.62) | 10.433962 (0.68) | 9.571429 (0.57) | 10.592593 (0.61) | 9.760417 (0.63)
  Session 3: number analyzed (Participants) | 23 | 41 | 28 | 38 | 35 | 51
  Session 3 | 7.782609 (0.47) | 9.292683 (0.60) | 10.285714 (0.57) | 8.526316 (0.53) | 10.171429 (0.58) | 8.745098 (0.65)
  Session 4: number analyzed (Participants) | 16 | 35 | 20 | 35 | 21 | 32
  Session 4 | 8.750000 (0.48) | 8.514286 (0.57) | 10.600000 (0.47) | 7.771429 (0.62) | 10.142857 (0.49) | 8.406250 (0.50)
  Session 5: number analyzed (Participants) | 15 | 28 | 17 | 30 | 15 | 26
  Session 5 | 9.066667 (0.45) | 8.535714 (0.59) | 10.058824 (0.64) | 7.666667 (0.53) | 8.071429 (0.57) | 8.115385 (0.52)
  Session 6: number analyzed (Participants) | 14 | 28 | 15 | 24 | 14 | 22
  Session 6 | 7.928571 (0.43) | 8.407407 (0.53) | 9.200000 (0.58) | 8.391304 (0.45) | 8.714286 (0.50) | 8.500000 (0.58)
  Session 7: number analyzed (Participants) | 10 | 27 | 11 | 23 | 14 | 19
  Session 7 | 7.222222 (0.54) | 8.285714 (0.54) | 8.818182 (0.49) | 7.681818 (0.73) | 8.384615 (0.46) | 7.631579 (0.52)
  Session 8: number analyzed (Participants) | 9 | 23 | 11 | 22 | 13 | 14
  Session 8 | 9.200000 (0.30) | 9.521739 (0.57) | 11.454545 (0.68) | 8.041667 (0.42) | 7.400000 (0.47) | 7.357143 (0.50)
  2-month Follow-up: number analyzed (Participants) | 1 | 5 | 3 | 6 | 7 | 2
  2-month Follow-up | 3.000000 (0.55) | 7.400000 (0.53) | 11.333333 (0.45) | 8.333333 (0.58) | 8.000000 (0.50) | 6.000000 (0.63)
Statistical Analysis 1: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, Likelihood Ratio Tests — =Positive~No-training, 0.130=Positive~50/50 training, 0.269=50/50~No-training Alpha = .05; 2=Positive~No-training, 2=Positive~50/50 training, 2=50/50~No-training; Mean Difference (Net) = 11.551 — =Positive~No-training, 4.075=Positive~50/50 training, 2.630=50/50~No-training
Statistical Analysis 2: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.140, Likelihood Ratio Tests — Alpha = .05; 2=df Neutral~Anxiety prime; Mean Difference (Net) = 3.933
Statistical Analysis 3: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.049, Likelihood Ratio Tests — =No-train+Neut~Pos+Anx,0.049=No-train+Neut~Pos+Neut,Positive(all)~No-train+Anx≥0.198,50/50(all)~No-train+Anx≥0.104,0.014=No-train+Neut~50/50+Neut,0.627=No-train+Neut~50/50+Anx,0.021=Pos+Anx~50/50+Anx,0.764=Pos+Anx~50/50+Neut,Pos+Neut~50/50(all)≥0.067; 2=all df; Mean Difference (Net) = 6.018 — =No-train+Neut~Pos+Anx,6.041=No-train+Neut~Pos+Neut,Positive(all)~No-train+Anx≤3.240,50/50(all)~No-train+Anx≤4.534,8.525=No-train+Neut~50/50+Neut,0.933=No-train+Neut~50/50+Anx,7.686=Pos+Anx~50/50+Anx,0.537=Pos+Anx~50/50+Neut,Pos+Neut~50/50(all)≤5.395

3. Primary Outcome: Change in Recognition Ratings (Negative Interpretation Bias)
Description: To measure interpretation bias, participants will read ambiguous scenarios with titles, after which they will see the titles of each scenario, followed by 2 disambiguated interpretations of the scenario: 1 positive and 1 negative. Participants will rate each disambiguated interpretation based on how similar in meaning it is to the original scenario on a 4-point scale ranging from 1 to 4. The mean of the negative, threat-related ratings index negative interpretation bias. Higher scores represent a more negative interpretation bias.
Time Frame: as for outcome 1
Population: Due to attrition, the number of participants differs at each session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 111 | 141 | 121 | 144 | 136 | 154
score on a scale
  Baseline: number analyzed (Participants) | 110 | 140 | 120 | 143 | 110 | 125
  Baseline | 1.66 (0.94) | 1.70 (0.89) | 1.75 (0.87) | 1.74 (0.92) | 1.77 (0.84) | 1.77 (0.88)
  Session 3: number analyzed (Participants) | 23 | 41 | 25 | 40 | 32 | 47
  Session 3 | 1.21 (0.83) | 1.38 (0.79) | 1.74 (0.85) | 1.68 (0.92) | 1.85 (0.86) | 1.54 (0.84)
  Session 6: number analyzed (Participants) | 15 | 28 | 15 | 22 | 13 | 25
  Session 6 | 1.04 (0.73) | 1.18 (0.76) | 1.88 (0.86) | 1.67 (0.90) | 1.78 (0.76) | 1.52 (0.83)
  Session 8: number analyzed (Participants) | 9 | 22 | 10 | 20 | 12 | 14
  Session 8 | 1.20 (0.73) | 1.30 (0.72) | 1.51 (0.99) | 1.58 (0.90) | 1.83 (0.68) | 1.50 (0.77)
  2-month Follow-up: number analyzed (Participants) | 2 | 4 | 4 | 5 | 7 | 2
  2-month Follow-up | 1.17 (0.97) | 1.25 (0.70) | 1.67 (0.59) | 1.78 (0.71) | 1.73 (0.67) | 0.78 (0.26)
Statistical Analysis 1: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Likelihood Ratio Tests — =Positive~No-training, Positive~50/50 training<0.001, 0.124=50/50~No-training Alpha = .05; 2=df Positive~No-training, 2=df Positive~50/50 training, 2=df 50/50~No-training; Mean Difference (Net) = 17.420 — =Positive~No-training, 31.921=Positive~50/50 training, 4.175=50/50~No-training
Statistical Analysis 2: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.728, Likelihood Ratio Tests — =Neutral~Anxiety prime Alpha = .05; 2=df Neutral~Anxiety prime; Mean Difference (Net) = 0.634 — =Neutral~Anxiety prime
Statistical Analysis 3: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, Likelihood Ratio Tests — =Pos+Anx~No-train+Neut, 0.026=Pos+Anx~No-train+Anx, 0.002=Pos+Neut~No-train+Neut, 0.091=Pos+Neut~No-train+Anx, 50/50(all)~No-train(all)≥ 0.081, Positive(all)~50/50(all)< 0.001; 2=all df; Mean Difference (Net) = 15.034 — =Pos+Anx~No-train+Neut, 7.306=Pos+Anx~No-train+Anx, 12.672=Pos+Neut~No-train+Neut, 4.802=Pos+Neut~No-train+Anx, 50/50(all)~No-train(all)≤5.037, Positive(all)~50/50(all)≥16.239

4. Primary Outcome: Change in Brief Bodily Sensations Interpretations Questionnaire
Description: The Brief Bodily Sensation Interpretation Questionnaire (BBSIQ; Clark et al., 1997) was administered as a more independent, additional measure of interpretation bias. In the BBSIQ, participants are presented with fourteen ambiguous events related to physical (e.g., feeling lightheaded) or external (e.g., smelling smoke, social situations) concerns, along with three possible explanations for each ambiguous event (one negative, and two neutral or positive explanations). Participants rated the extent to which they believed each explanation for why the ambiguous event occurred on a Likert scale from 0 ("not at all likely") to 4 ("extremely likely"). Typically, the BBSIQ is administered on an eight-point Likert scale, but a 0-4 scale was used to align with other rating scales in the study. Negative interpretation bias score was computed by averaging the likelihood ratings for all negative explanations (following Steinman & Teachman, 2010, 2015).
Time Frame: as for outcome 1
Population: Due to attrition, the number of participants differs at each session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 111 | 141 | 121 | 144 | 136 | 154
units on a scale
  Baseline: number analyzed (Participants) | 111 | 141 | 121 | 140 | 133 | 150
  Baseline | 1.81 (1.15) | 1.83 (1.16) | 1.93 (1.17) | 1.91 (1.16) | 1.90 (1.13) | 1.85 (1.12)
  Session 3: number analyzed (Participants) | 23 | 42 | 25 | 39 | 31 | 45
  Session 3 | 1.82 (1.16) | 1.82 (1.17) | 1.80 (1.04) | 1.94 (1.14) | 1.86 (1.11) | 1.77 (1.03)
  Session 6: number analyzed (Participants) | 13 | 28 | 15 | 22 | 13 | 24
  Session 6 | 1.66 (1.09) | 1.85 (1.16) | 1.94 (1.13) | 1.94 (1.27) | 1.92 (1.22) | 1.90 (1.08)
  Session 8: number analyzed (Participants) | 9 | 22 | 10 | 20 | 12 | 15
  Session 8 | 1.58 (1.14) | 1.78 (1.16) | 1.90 (1.15) | 1.85 (1.24) | 1.87 (1.07) | 1.82 (1.17)
  2-month Follow-up: number analyzed (Participants) | 2 | 5 | 4 | 5 | 7 | 2
  2-month Follow-up | 1.68 (1.33) | 1.59 (0.80) | 2.04 (1.06) | 1.98 (1.30) | 2.13 (1.22) | 1.25 (1.04)
Statistical Analysis 1: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Likelihood Ratio Tests — =Positive~No-training, Positive~50/50 training< 0.001, 0.100=50/50~No-training Alpha = .05; 2=df Positive~No-training, 2=df Positive~50/50 training, 2=df 50/50~No-training; Mean Difference (Net) = 13.924 — =Positive~No-training, 15.288=Positive~50/50 training, 4.605=50/50~No-training
Statistical Analysis 2: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.135, Likelihood Ratio Tests — =Neutral~Anxiety prime Alpha = .05; 2=df Neutral~Anxiety prime; Mean Difference (Net) = 4.011 — =Neutral~Anxiety prime
Statistical Analysis 3: Comparison: Positive Training+Anxious Imagery Prime vs Positive Training+Neutral Imagery Prime vs 50/50 Training+Anxious Imagery Prime vs 50/50 Training+Neutral Imagery Prime vs No Scenario+Anxious Imagery Prime vs No Scenario+Neutral Imagery Prime; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.009, Likelihood Ratio Tests — =Pos+Anx~No-train+Neut, Pos+Anx~No-train+Anx<0.048, Pos+Neut~No-train+Neut<0.001, 0.055=Pos+Neut~No-train+Anx, 50/50(all)~No-train+Anx≥0.139, 0.034=No-train+Neut~50/50+Neut, 0.340=No-train+Neut~50/50+Anx, Pos(all)~50/50(all)≥ 0.087; 2=all df; Mean Difference (Net) = 9.402 — =Pos+Anx~No-train+Neut, 6.076=Pos+Anx~No-train+Anx, 14.525=Pos+Neut~No-train+Neut, 5.811=Pos+Neut~No-train+Anx, 50/50(all)~No-train+Anx≤3.950, 6.770=No-train+Neut~50/50+Neut, 2.158=No-train+Neut~50/50+Anx, Pos(all)~50/50(all)≤4.876

5. Secondary Outcome: Multi-Session User Experience Questionnaire
Description: This questionnaire assesses users' opinions about the intervention. Participants could select from options "Not at all=0, Slightly=1, Somewhat=2, Mostly=3, Very=4, Decline to answer=5" for questions 1-13 as well as 15 and 16 (examples listed below); question 14 asked "This training program was 8 sessions. How many sessions do you think would have been ideal?" with an open ended response box, which we will not include in the means and SDs. We will recode "Decline to answer=5" as NA. Higher scores on this scale indicate more positive experiences with the program in general across questions, from 0-4.
  1. How helpful did you find the web program for reducing your anxiety?
  2. How much did the web program improve your overall quality of life?
  3. How much did the web program help improve your overall mood (e.g., feeling happier)?
  4. How likely would you be to recommend this web program to others with similar anxiety difficulties?
  5. How easy was the web program to use?
Time Frame: At 2-month follow-up
Population: Due to attrition, the number of participants differs at from the overall number in the participant flow, as user experience was only assessed at follow-up, during which we did not receive responses from a majority of participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 6 | 2
score on a scale | 2.54 (1.05) | 2.31 (1.36) | 2.66 (1.05) | 2.74 (1.03) | 2.81 (1.33) | 2.21 (1.09)

6. Secondary Outcome: Impact of Anxious Imagery Prime (Change Over Time is Exploratory But Should Show Anxious/Neutral Prime Differences; e.g., in Subjective Distress)
Description: Following the anxious or neutral imagery prime, participants reported on the questions provided. Minimum score = 3; maximum score =115. Higher scores indicate more vividness and anxiety following the anxious imagery prime.
  How vividly did you imagine the situation?
  1=Not at all vivid 2=Somewhat vivid 3=Moderately vivid 4=Very vivid 5=Totally vivid
  How anxious did you feel (at the highest level of anxiety) as you completed the imagery task? (using a 0-100 slider with the following anchors marked) 0=Not at all anxious, 50= Moderately anxious, 100=Totally anxious
  How likely is it that this situation will turn out well vs. turn out badly? 1=Very likely to turn out well, 2=Somewhat likely to turn out well, 3=Neutral, 4= Somewhat likely to turn out badly, 5= Very likely to turn out badly
  If this situation did turn out badly, how well or badly would you be able to handle it?
  1=Very well, 2=Somewhat well, 3=Neutral, 4=Somewhat badly, 5=Very badly
Time Frame: After sessions 1,2,3,4,5,6,7,8 (sessions will be spaced ~3-4 days apart). Measure will be completed following that day's imagery prime (which immediately precedes the training session).
Population: Due to attrition, the number of participants differs at each session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 111 | 141 | 121 | 144 | 136 | 154
score on a scale
  Session 1: number analyzed (Participants) | 74 | 87 | 76 | 86 | 93 | 103
  Session 1 | 18.73311 (30.59704) | 7.899425 (11.26371) | 18.77632 (30.67108) | 7.927326 (11.675453) | 18.57796 (30.46432) | 8.783981 (13.011083)
  Session 2: number analyzed (Participants) | 22 | 42 | 31 | 43 | 45 | 53
  Session 2 | 18.17045 (29.38720) | 7.154762 (10.01027) | 18.62903 (30.21894) | 6.808140 (9.383420) | 19.16111 (31.42217) | 6.867925 (9.533016)
  Session 3: number analyzed (Participants) | 14 | 32 | 20 | 28 | 24 | 38
  Session 3 | 17.76786 (28.40848) | 8.500000 (12.48014) | 18.68750 (30.42976) | 8.821429 (13.216355) | 19.04167 (31.10353) | 7.986842 (11.633403)
  Session 4: number analyzed (Participants) | 9 | 27 | 15 | 24 | 16 | 22
  Session 4 | 18.55556 (30.30694) | 7.879630 (11.37995) | 16.55000 (26.40416) | 8.375000 (12.900746) | 16.89062 (27.09552) | 8.556818 (12.628915)
  Session 5: number analyzed (Participants) | 6 | 22 | 14 | 20 | 12 | 17
  Session 5 | 19.16667 (30.67189) | 7.784091 (11.31204) | 17.87500 (28.95789) | 8.050000 (12.239715) | 14.39583 (22.71050) | 7.411765 (10.369064)
  Session 6: number analyzed (Participants) | 6 | 20 | 13 | 13 | 10 | 15
  Session 6 | 21.00000 (34.45232) | 7.637500 (11.05529) | 18.76923 (30.67833) | 8.307692 (12.367694) | 17.75000 (28.83588) | 8.050000 (11.665366)
  Session 7: number analyzed (Participants) | 4 | 17 | 11 | 13 | 10 | 12
  Session 7 | 16.75000 (27.00975) | 8.308824 (12.36007) | 17.79545 (28.39446) | 7.250000 (10.811497) | 17.27500 (27.77881) | 7.437500 (10.966967)
  Session 8: number analyzed (Participants) | 4 | 14 | 8 | 10 | 9 | 9
  Session 8 | 18.00000 (28.50996) | 10.017857 (15.63498) | 18.96875 (31.28617) | 5.725000 (8.042796) | 14.61111 (23.71496) | 7.083333 (10.676861)

7. Secondary Outcome: Change in Depression, Anxiety, Stress Scales-Short Form: Anxiety Subscale
Description: While we use the OASIS as a primary measure of anxiety symptom severity, we are using the DASS-AS (Lovibond & Lovibond, 1995) as another 7-item measure of anxiety symptoms. Higher scores indicate more severe anxiety symptoms. Minimum score = 0; maximum score = 21.
  0 = Did not apply to me at all
  1. = Applied to me to some degree, or some of the time
  2. = Applied to me to a considerable degree, or a good part of time
  3. = Applied to me very much, or most of the time
  Qs:
  1. I was aware of dryness of my mouth.
  2. I experienced breathing difficulty (e.g., excessively rapid breathing, breathlessness in the absence of physical exertion).
  3. I experienced trembling (e.g., in the hands).
  4. I was worried about situations in which I might panic and make a fool of myself.
  5. I felt I was close to panic.
  6. I was aware of the action of my heart in the absence of physical exertion (e.g., sense of heart rate increase, heart missing a beat).
  7. I felt scared without any good reason.
Time Frame: Baseline, after session 8 (~4 weeks after baseline) & at 2-month follow-up.
Population: Due to attrition, the number of participants differs at each session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 111 | 141 | 121 | 144 | 136 | 152
score on a scale
  Baseline | 22.4 (7.92) | 22.64 (7.91) | 24.7 (8.0) | 22.7 (7.93) | 23.84 (9.80) | 22.48 (7.94)
  Session 8: number analyzed (Participants) | 10 | 22 | 10 | 19 | 11 | 12
  Session 8 | 14.4 (9.11) | 14.3 (9.07) | 19.8 (9.20) | 11.37 (9.17) | 16.36 (9.10) | 14.17 (9.10)
  2-month Follow-up: number analyzed (Participants) | 2 | 5 | 4 | 6 | 6 | 2
  2-month Follow-up | 13 (9.72) | 15.6 (9.54) | 19.0 (9.60) | 10.67 (9.60) | 9.67 (9.29) | 14 (9.29)

8. Secondary Outcome: Change in Quality of Life Scale
Description: The Quality of Life Scale (Flanagan, 1978) is a 16-item questionnaire chosen to evaluate change in quality of life in five domains: recreation, relationships, well-being, personal fulfillment and development, and social activities. Higher scores indicate more positive feelings about quality of life/more satisfaction. Minimum score = 16; maximum score = 80.
  The question asks "How satisfied are you with..." with each of the following options as separate questions: material, health, relationships, children, spouse, friend, helping, participating, learning, understanding, work, expression, socializing, reading, recreation, independence (just providing a key word for purposes of description, but questions include a full statement such as "Material comforts home, food, conveniences, financial security " for material).
  Response options range from Completely unsatisfied=1, Somewhat unsatisfied=2, Mixed=3, Somewhat satisfied=4, Completely satisfied=5.
Time Frame: as for outcome 1
Population: Number of participants varies by session due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
Number analyzed (Participants) | 111 | 141 | 120 | 144 | 135 | 149
score on a scale
  Baseline | 3.196459 (1.0354441) | 3.106346 (1.0543742) | 3.081101 (1.0750755) | 3.169298 (1.0052069) | 3.157229 (1.0582803) | 3.283237 (1.0084809)
  Session 3: number analyzed (Participants) | 23 | 42 | 25 | 39 | 31 | 45
  Session 3 | 3.182143 (0.8987590) | 3.088767 (0.9424159) | 3.123667 (1.0305259) | 3.314192 (0.9043169) | 2.985270 (1.0139484) | 3.275440 (0.8989526)
  2Session 6: number analyzed (Participants) | 13 | 28 | 15 | 23 | 13 | 24
  2Session 6 | 2.975962 (0.8749633) | 3.089638 (0.9243989) | 3.166667 (1.0418765) | 3.409006 (0.9131546) | 2.955463 (0.9939990) | 3.443031 (0.8065981)
  Session 8: number analyzed (Participants) | 9 | 22 | 10 | 20 | 12 | 15
  Session 8 | 2.957341 (0.9889570) | 2.939854 (0.9254448) | 3.006250 (1.0276903) | 3.479613 (0.9089624) | 3.114583 (1.0242228) | 3.515278 (0.7620035)
  2-month Follow-up: number analyzed (Participants) | 2 | 5 | 4 | 5 | 7 | 2
  2-month Follow-up | 3.625000 (0.9350209) | 3.775000 (0.6580935) | 3.232292 (0.9395024) | 3.675000 (0.8625170) | 2.899150 (0.9038532) | 4.080357 (0.6680277)

ADVERSE EVENTS:
Time Frame: Adverse event data was monitored throughout the study, through study completion (during the weeks of active study sessions and at 2 month follow-up).
Description: Adverse events were investigated by researchers regularly.
Arm/Group | Positive Training+Anxious Imagery Prime | Positive Training+Neutral Imagery Prime | 50/50 Training+Anxious Imagery Prime | 50/50 Training+Neutral Imagery Prime | No Scenario+Anxious Imagery Prime | No Scenario+Neutral Imagery Prime
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/141 | 0/121 | 0/144 | 0/136 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/141 | 0/121 | 0/144 | 0/136 | 0/154
Other Adverse Events (participants affected / at risk) | 0/111 | 0/141 | 0/121 | 0/144 | 0/136 | 0/154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT02382003/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02382003/ICF_001.pdf